CLINICAL TRIAL: NCT06033937
Title: Comparison of the Effect of Device Closure in Alleviating Migraine With Patent Foramen Oval: COMPETE Cohort Study
Brief Title: COMPETE Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Principal investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2022-1758-2
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: PFO - Patent Foramen Ovale; Migraine
MeSH Terms: conditions — Foramen Ovale, Patent; Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Migraine Medication Group
- PFO Occlusion Group
  Interventions: Device: PFO occlusion

INTERVENTIONS:
Device: PFO occlusion — Patients in PFO occlusion group received PFO closure using devices.
  Groups: PFO Occlusion Group

SUMMARY:
Migraine attacks are episodic disorder that affects approximately 12% of the population, and studies have shown that 41-48% of migraineurs have a combination of patent foramen ovale (PFO). Clinical Observational studies have been linking PFO occlusion with the effectiveness in improving migraine symptoms and reducing the frequency of attacks. However, several RCTs have shown negative primary results, making it unclear whether PFO occlusion is effective in treating migraine. Our study is a multi-center cohort study aiming to find the correlation between PFO closure and migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 ；
2. Diagnosed migraine by ICHD-3
3. History of migraine longer than 1 year, and symptoms severely disturbing daily life.
4. TCD/TTE/TEE diagnosed patent foramen ovale with right to left shunt
5. Willing to participant and agree to follow-ups
6. Received at least three different types of migraine preventive drugs, the responder rate of previous therapy did not receive 50%.

Exclusion Criteria:

1. Migraine caused by other reason
2. Had TIA/stroke history
3. With contraindication or hypersensitive to anti-platelet or anticoagulation drugs.
4. With contraindication to PFO occlusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with PFO and migraine who met the eligibility criteria are recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Responder rate | From baseline period to 12-month treatment period
  Defined as a 50% reduction from the monthly number of migraine attacks during the baseline phase to the monthly number of migraine attacks during the treatment phase.

SECONDARY OUTCOMES:
Migraine days change per month | From baseline period to 12-month treatment period
  Change in the mean number of migraine days from baseline to treatment phase.
Number of migraine attacks change per month | From baseline period to 12-month treatment period
  Change in the mean number of migraine attacks from baseline to treatment phase.
Percentage of complete migraine cessation | From baseline period to 12-month treatment period
  Participants experienced complete migraine attacks cessation after treatment phase as compared to baseline phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China